CLINICAL TRIAL: NCT04511208
Title: Cooling Vest May Reduce Heat Stress, Improve Thermal Comfort, and Preserve Cognitive Performance of Surgeons While Performing Surgery
Brief Title: Cooling Vest May Reduce Heat Stress During Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20-214
Record Dates: First submitted 2020-07-19; First posted 2020-08-13 (Actual); Results first posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Body Temperature Changes
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Cooling vest, then without cooling vest, then without cooling vest, then cooling vest (ABBA) (Experimental): Surgeons first performed one surgery with the cooling vest. On another day, they then performed one surgery without the cooling vest. Then on another day, they performed another surgery without the cooling vest. Then they finally performed one surgery with the cooling vest.
  Interventions: Device: Cooling Vest; Device: Without cooling vest
- Without cooling vest, then cooling vest, then cooling vest, then without cooling vest (BAAB) (Experimental): Surgeons first performed one surgery without the cooling vest. On another day, they then performed one surgery with the cooling vest. Then on another day, they performed another surgery with the cooling vest. Then they finally performed one surgery without the cooling vest.
  Interventions: Device: Cooling Vest; Device: Without cooling vest
- Cooling vest, then cooling vest, then without cooling vest, then without cooling vest (AABB) (Experimental): Surgeons first performed one surgery with the cooling vest. On another day, they then performed another surgery with the cooling vest. Then on another day, they performed one surgery without the cooling vest. Then they finally performed another surgery without the cooling vest.
  Interventions: Device: Cooling Vest; Device: Without cooling vest
- Without cooling vest, then without cooling vest, then cooling vest, then cooling vest (BBAA) (Experimental): Surgeons first performed one surgery without the cooling vest. On another day, they then performed another surgery without the cooling vest. Then on another day, they performed one surgery with the cooling vest. Then they finally performed another surgery with the cooling vest.
  Interventions: Device: Cooling Vest; Device: Without cooling vest

INTERVENTIONS:
Device: Cooling Vest — Evaluate that wearing a cooling vest during surgery reduces surgeons' mean-body temperature and preserves their cognitive performance.
Device: Without cooling vest — Evaluate surgeons' mean-body temperature and cognitive performance without cooling vest.

SUMMARY:
The investigators will propose a randomized cross-over trial using a uniform and strongly balanced 4-period design in which will include four operations for each surgeon. Surgeons will be randomized to 1 of 4 sequences: ABBA, BAAB, AABB or BBAA. The design is "uniform" in that each treatment appears the same number of times within each sequence (uniform within sequence) and if each treatment appears the same number of times within each period (uniform within each period). It is strongly balanced with respect to first-order carryover effects because each treatment precedes every other treatment, including itself, the same number of times

DETAILED DESCRIPTION:
The subjects will be randomly assigned to use either the CoolSource™ cooling vest (worn between scrubs) and a conventional surgical gown for each of 4 surgeries. Sequence of treatments within the subjects will be randomized (ABBA, BAAB, AABB or BBAA), and determined using the PLAN procedure in SAS, such that each surgeon will wear vest and non-vest twice. The sequencing will not be shared with any study personnel. Allocation for each case will be concealed with a web-based system that will be accessed only shortly before surgery.

The investigators will target an ambient temperature of 21°C ± 1°C, and try to maintain the same temperature of each of the four study cases for each surgeon. The CoolSource vest holds six reusable cooling packs located bilaterally on the shoulders, angled flank along the base of the rib cage, and along each side of the spine, mid-back. The vest will be donned over hospital-issued scrubs after all temperature sensing devices have been applied and before surgical hand scrubbing. The subjects will wear the vest throughout surgery, and for a few additional minutes while postoperative assessments are made (details below).

The weight of the disposable cooling vest is 1 kg which is evenly distributed over both shoulders. The cooling packs have an insulated cover to reduce condensation or sweating while seated inside the vest pocket. The flexible frozen reusable cooling packs will be inserted into each of the six pockets and the vest belt will be tied to hold the cooling packs securely. The disposable cooling vests will be discarded after each case, and the cooling packs returned to a freezer.

ELIGIBILITY:
Inclusion Criteria:

* Surgeons who perform elective major orthopedic surgery such as total hip and knee arthroplasties scheduled for 90 to 150 minutes at the Cleveland Clinic Main Campus.
* Orthopedic surgeons ages of 25-65 years old, as body temperatures may be lower and less stable in the elderly (Waalen & Buxbaum, 2011), who operate frequently enough to participate in four cross-over cases.
* Surgical helmet system is consistently worn for each of the surgeon's four cases, if used in the first case.

Exclusion Criteria:

* Surgical cases that require surgeons to sit on stools during the procedure, which may impact temperature and energy expenditure.
* - Surgeons who report having a recent illness within 24 hours prior to the surgery, symptoms producing a febrile condition;
* Surgeons who worked the previous evening.
* Surgeons who wear lead X-ray gowns.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2022-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share data on a collaborative basis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of the primary paper.
Access Criteria: Collaborative proposal approved by the trial Executive Committee. Data use agreement will be required. Address requests to Daniel Sessler at DS@CCF.org.

REFERENCES:
- [Derived] Byrne JE, Rodriguez-Patarroyo FA, Mascha EJ, Han Y, Bravo M, Bloomfield MR, Rao SM, Sessler DI. Cooling vest improves surgeons' thermal comfort without affecting cognitive performance: a randomised cross-over trial. Occup Environ Med. 2023 Jun;80(6):339-345. doi: 10.1136/oemed-2022-108457. Epub 2023 May 4. PMID 37142418

RESULTS

PARTICIPANT FLOW:
Period: First Surgery
Arm/Group | Cooling Vest, Then Without Cooling Vest, Then Without Cooling Vest, Then Cooling Vest (ABBA) | Without Cooling Vest, Then Cooling Vest, Then Cooling Vest, Then Without Cooling Vest (BAAB) | Cooling Vest, Then Cooling Vest, Then Without Cooling Vest, Then Without Cooling Vest (AABB) | Without Cooling Vest, Then Without Cooling Vest, Then Cooling Vest, Then Cooling Vest (BBAA)
Started | 8 | 7 | 8 | 7
Completed | 8 | 7 | 8 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Second Surgery
Arm/Group | Cooling Vest, Then Without Cooling Vest, Then Without Cooling Vest, Then Cooling Vest (ABBA) | Without Cooling Vest, Then Cooling Vest, Then Cooling Vest, Then Without Cooling Vest (BAAB) | Cooling Vest, Then Cooling Vest, Then Without Cooling Vest, Then Without Cooling Vest (AABB) | Without Cooling Vest, Then Without Cooling Vest, Then Cooling Vest, Then Cooling Vest (BBAA)
Started | 8 | 7 | 8 | 7
Completed | 8 | 7 | 8 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Third Surgery
Arm/Group | Cooling Vest, Then Without Cooling Vest, Then Without Cooling Vest, Then Cooling Vest (ABBA) | Without Cooling Vest, Then Cooling Vest, Then Cooling Vest, Then Without Cooling Vest (BAAB) | Cooling Vest, Then Cooling Vest, Then Without Cooling Vest, Then Without Cooling Vest (AABB) | Without Cooling Vest, Then Without Cooling Vest, Then Cooling Vest, Then Cooling Vest (BBAA)
Started | 8 | 7 | 8 | 7
Completed | 8 | 7 | 8 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Forth Surgery
Arm/Group | Cooling Vest, Then Without Cooling Vest, Then Without Cooling Vest, Then Cooling Vest (ABBA) | Without Cooling Vest, Then Cooling Vest, Then Cooling Vest, Then Without Cooling Vest (BAAB) | Cooling Vest, Then Cooling Vest, Then Without Cooling Vest, Then Without Cooling Vest (AABB) | Without Cooling Vest, Then Without Cooling Vest, Then Cooling Vest, Then Cooling Vest (BBAA)
Started | 8 | 7 | 8 | 7
Completed | 8 | 7 | 8 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants were randomized to receive all interventions
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 26
  Asian | 2
  Black/African American | 1
  Hispanic/Latino | 1
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 26 [25 to 28]
Height [Median (Inter-Quartile Range); unit: cm] | 181 [178 to 183]
Weight [Median (Inter-Quartile Range); unit: kg] | 85 [82 to 98]

OUTCOME MEASURES:

1. Primary Outcome: Self-rated Thermal Comfort.
Description: Immediately after surgery, while still gowned, surgeons will rate their thermal comfort on a 0-10 Likert scale, with 0 representing extreme cold, 5 being thermal comfort, and 10 representing extreme heat. Two points on the 11-point Likert scale will be considered a clinically important difference.
Time Frame: Immediately after surgery, within 10 minutes
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Surgeries
Groups:
- Cooling Vest: Evaluate surgeons' self-rated thermal comfort using the cooling Ice vest during prolonged and strenuous surgery
  Cooling Vest: Evaluate that wearing a cooling vest during surgery reduces surgeons' mean-body temperature and preserves their cognitive performance.
- Without Cooling Vest: Evaluate surgeons' self-rated thermal comfort without using the Cooling Ice Vest during prolonged and strenuous surgery
  Cooling Vest: Evaluate that wearing a cooling vest during surgery reduces surgeons' mean-body temperature and preserves their cognitive performance.
  Control Group without cooling vest: Evaluate surgeons' mean-body temperature and cognitive performance without cooling vest.
Arm/Group | Cooling Vest | Without Cooling Vest
Number analyzed (Participants) | 30 | 30
Number analyzed (Surgeries) | 60 | 60
score on a scale | 4.4 (0.19) | 6.6 (0.19)
Statistical Analysis 1: Comparison: Cooling Vest vs Without Cooling Vest; Test type: Superiority; p < 0.001, Repeated measures linear model; Difference in means = -2.2, 95% CI 2-sided [-2.7 to -1.7]

2. Secondary Outcome: Mean Core Temperature.
Description: The first secondary outcome will be the mean core temperature for a case, calculated as the time-weighted average over the taken measurements. The surgeon's core body temperature will be monitored by a validated wireless wearable iThermonitor WT701 biosensor which estimates core temperature within ±0.5⁰C (Pei et al., 2018). The sensor will be applied to the surgeon's right axilla 15-20 minutes prior to the surgical hand scrub performed at the start of surgery and secured with an adhesive cover. A small patch of axillary hair will be clipped or shaved as necessary.
Time Frame: the sensor will be worn for a total of 90 minutes
Measure: Mean (Standard Error); unit: ℃
Units Other Than Participants: Surgeries
Arm/Group | Cooling Vest | Without Cooling Vest
Number analyzed (Participants) | 30 | 30
Number analyzed (Surgeries) | 60 | 60
℃ | 32.9 (0.09) | 33.2 (0.09)
Statistical Analysis 1: Comparison: Cooling Vest vs Without Cooling Vest; Test type: Superiority; p = 0.006, Repeated measures linear model; Difference in means = -0.26, 95% CI 2-sided [-0.44 to -0.08]

3. Secondary Outcome: Mean Skin Temperature
Description: The second secondary outcome will be the mean skin temperature for a case, calculated as the time-weighted average over the taken measurements. Mean skin temperature will be estimated from skin temperature from the back of the upper chest, deltoid arm, thigh, and calf using the formula [MSTR = 0.3 chest + 0.3 arm + 0.2 thigh + 0.2 leg or 0.3(chest + arm) + 0.2(thigh + 0.2 leg)] (Ramanathan, 1964). Skin temperature will be continuously measured using wireless patches, TempTraq, which meet professional accuracy standards for digital thermometers (ASTM E1112-00). The sensors will remain affixed with adhesive dressing on the surgeon's body surface throughout surgery and approximately 10 minutes required for post-operative testing.
Time Frame: the sensor will be worn for a total of 90 minutes
Measure: Mean (Standard Error); unit: ℃
Units Other Than Participants: Surgeries
Arm/Group | Cooling Vest | Without Cooling Vest
Number analyzed (Participants) | 30 | 30
Number analyzed (Surgeries) | 60 | 60
℃ | 36.1 (0.13) | 36.3 (0.13)
Statistical Analysis 1: Comparison: Cooling Vest vs Without Cooling Vest; Test type: Superiority; p = 0.046, Repeated measures linear model; Difference in means = -0.23, 95% CI 2-sided [-0.45 to -0.005]

4. Secondary Outcome: Surgeons' Cognitive Performance, Measured With the C3B Battery.
Description: Surgeons' cognitive performance was assessed with the Cleveland Clinic Cognitive Battery (C3B, Cleveland, OH), a ten-minute-long self-administered computer tablet program that tests visual memory (episodic learning and delayed memory, range 0 - 70) and processing speed (information processing speed and incidental memory, range 40 - 120). Testing will take place right after surgery with surgeons still gowned. The surgeons will sit with the iPad touch screen placed on a desk in front of them for approximately 10 minutes to complete the cognitive test.
Time Frame: Immediately after surgery, within 10 minutes
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Surgeries
Arm/Group | Cooling Vest | Without Cooling Vest
Number analyzed (Participants) | 30 | 30
Number analyzed (Surgeries) | 60 | 60
score on a scale
  C3B Processing Speed Test Score | 69.4 (0.82) | 69.4 (0.82)
  C3B Visual Memory Test Score | 58.3 (1.42) | 57.7 (1.41)
Statistical Analysis 1: Comparison: Cooling Vest vs Without Cooling Vest; C3B PST Score; Test type: Superiority; p = 0.955, Repeated measures linear model; Difference in means = -0.07, 95% CI 2-sided [-2.51 to 2.38]
Statistical Analysis 2: Comparison: Cooling Vest vs Without Cooling Vest; C3B VMT Score; Test type: Superiority; p = 0.686, Repeated measures linear model; Difference in means = 0.62, 95% CI 2-sided [-2.48 to 3.71]

5. Secondary Outcome: Surgeon' Perceived Ergonomic Workload Measured With the Borg Rating of Perceived Exertion (RPE) Scale.
Description: Immediately after surgery, while still gowned, surgeons will rate their perceived exertion on the Borg scale which ranges from 6 (no exertion) to 20 (maximal exertion).
Time Frame: Immediately after surgery, within 10 minutes
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: Surgeries
Arm/Group | Cooling Vest | Without Cooling Vest
Number analyzed (Participants) | 30 | 30
Number analyzed (Surgeries) | 60 | 60
score on a scale | 13 [11 to 13] | 13 [12 to 15]
Statistical Analysis 1: Comparison: Cooling Vest vs Without Cooling Vest; Test type: Superiority; p = 0.007, Generalized linear mixed effects model; Odds Ratio (OR) = 2.5, 95% CI 2-sided [1.28 to 4.68]
Statistical Analysis 2: Comparison: Cooling Vest vs Without Cooling Vest; Sensitivity analysis; Test type: Superiority; p = 0.009, Repeated measures linear model; Difference in means = -1.1, 95% CI 2-sided [-1.82 to -0.28]

6. Secondary Outcome: Surgeon' Perceived Fatigue Measured as 0 Representing Not Fatigued at All, 5 Moderately Fatigued, and 10 Total Fatigue & Exhaustion
Description: Perceived fatigue will be rated on a 0-10 ROF scale, with 0 representing not fatigued at all, 5 moderately fatigued, and 10 total fatigue & exhaustion. Two points difference on either scale will be considered a clinically important difference.
Time Frame: Immediately after surgery, within 10 minutes
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Surgeries
Arm/Group | Cooling Vest | Without Cooling Vest
Number analyzed (Participants) | 30 | 30
Number analyzed (Surgeries) | 60 | 60
score on a scale | 2.3 (0.26) | 3.3 (0.25)
Statistical Analysis 1: Comparison: Cooling Vest vs Without Cooling Vest; Test type: Superiority; p = 0.004, Repeated measures linear model; Difference in means = -1.06, 95% CI 2-sided [-1.75 to -0.38]

7. Secondary Outcome: Surgeons' Perception and Amount of Sweat-soaked Scrub Clothing.
Description: Immediately after surgery, while still gowned, surgeons' perception and amount of sweat-soaked scrub clothing will be rated using a Likert scale from 0 = "not wet at all" to 10 = "fully drenched."
Time Frame: Immediately after surgery, within 10 minutes
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Surgeries
Arm/Group | Cooling Vest | Without Cooling Vest
Number analyzed (Participants) | 30 | 30
Number analyzed (Surgeries) | 60 | 60
score on a scale | 1.4 (0.38) | 4.4 (0.38)
Statistical Analysis 1: Comparison: Cooling Vest vs Without Cooling Vest; Test type: Superiority; p < 0.001, Repeated measures linear model; Difference in means = -2.97, 95% CI 2-sided [-3.80 to -2.13]

ADVERSE EVENTS:
Time Frame: From the surgeons putting on the sterile surgical gown and the cooling vest to the time they remove the sterile surgical gown and the cooling vest after completing the postoperative assessments, with an average of 140 minutes.
Groups:
- Cooling Ice Vest: Evaluate surgeons' self-rated thermal comfort using the cooling Ice vest during prolonged and strenuous surgery
  Cooling Vest: Evaluate that wearing a cooling vest during surgery reduces surgeons' mean-body temperature and preserves their cognitive performance.
- Without Cooling Ice Vest: Evaluate surgeons' self-rated thermal comfort without using the Cooling Ice Vest during prolonged and strenuous surgery
  Cooling Vest: Evaluate that wearing a cooling vest during surgery reduces surgeons' mean-body temperature and preserves their cognitive performance.
  Control Group without cooling vest: Evaluate surgeons' mean-body temperature and cognitive performance without cooling vest.
Arm/Group | Cooling Ice Vest | Without Cooling Ice Vest
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT04511208/Prot_SAP_000.pdf